CLINICAL TRIAL: NCT01219816
Title: Phase II, Multicenter, Open Label, Prospective to Evaluate Efficacy and Tolerance of a Chemoimmunotherapy With HyperCVAD or Vincristine/Dexamethasone Plus the Anti-CD22 Monovlonal Antobody Epratuzumab for the Treatment of Adult Relapsed/Refractory CD22+ B-Acute Lymphoblastic Leukaemia Patients : CHEPRALL Study, a GRAALL Study.
Brief Title: Multi-centric Study
Acronym: CHEPRALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/10/05-O
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2016-11

CONDITIONS: B ALL; CD22+ Expression; Refractory B-ALL
Keywords: efficacy of Chemo-immunotherapy
MeSH Terms: interventions — epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients under 60 years (Experimental): Hyper CVAD regimen + Epratuzumab (Cyclophosphamide Vincristine Doxorubicin Dexamethasone)
  Interventions: Drug: Epratuzumab
- Patients older than 60 years or < =60 years (Experimental): Vincristine + Aracytine + Dexamethasone
  Interventions: Drug: Epratuzumab

INTERVENTIONS:
Drug: Epratuzumab — Combination of chemotherapy + Epratuzumab
  Arms: Patients under 60 years
Drug: Epratuzumab — Vincristine + Dexamethasone + Epratuzumab
  Arms: Patients older than 60 years or < =60 years

SUMMARY:
Patients with relapsed/refractory adult acute lymphoblastic leukemia (ALL)have a very dismal prognosis. In this case, allogeneic transplantation is the only curative treatment when patient have obtained a second complete remission (CR. In France, in patients younger than 60 years old,the HyperCVAD regimen used by the MDAnderson in Houston is generally applied. In older patients (>=60 years)or young patients <= 60 years no eligible for intense chemotherapy, a combination of vincristine + Dexamethasone is generally chosen in order to avoid too much toxicity but the result is worse in term of CR.

More than 90% of ALL with a B phenotype (2/3 of cases in adults)express the surface antigen CD22 on leukemic blasts which thus represents an interesting target for therapy. Epratuzumab is a humanized anti-CD22 antibody produced by Immunomedics, Inc, Morris Plain (New Jersey, USA). Epratuzumab has already shown efficacy in lymphoma patients. Only one study, including 15 children, has been published so far reporting the efficacy and the toxicity of Epratuzumab in the setting of ALL in monotherapy, one can observe 8 stable disease, 3 progressions and 4 partial responses. When combining chemotherapy and Epratuzumab, 9CR were observed with acceptable toxicity. Tolerance was acceptable.

The French GRAALL group proposes to test an age-adapted combination of chemotherapy + Epratuzumab, in refractory/relapses CD22+ B ALL patients in order to improve their prognosis, in term of CR, survival and of number of patients eligible for allograft.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* B-ALL (OMs) with >= 20 % of blasts in bone marrow
* CD22+ expression >= 30% of the blast population
* Refractory B-ALL defined by treatment failure after 2 successive courses of induction therapy or relapse < 6 months after first CR
* First relapse of B-ALL
* Second relapse or beyond
* Performance status 0-2
* Creatinine clearance >= 50 ml/min (Cockroft formula)
* Serum bilirubine <= 30 µmom/l
* Written informed consent

Exclusion Criteria:

* T-ALL
* Meningeal involvement
* CD22 expression on tumor cells or < 30%
* HIV positive
* Active Hepatitis B or C
* Left ventricular ejection fraction < 50% in patients <60 years
* Contra-indication to Epratuzumab
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 5 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Participation at the same time in another study in which investigational drugs are used
* Absence of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
complete response rate (CR and CRp)

SECONDARY OUTCOMES:
Overall response rate (ORR)(CR, CRp and PR)
Overall survival
Disease free survival
CD22 expression after Epratuzumab
Safety and tolerance of Epratuzumab in combination with chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Patrice CHEVALLIER, MD, Principal Investigator — Nantes University Hospital
Locations (11):
- France (11):
  - Angers University Hospital, Angers
  - University Hospital, Caen
  - HEnri Mondor Hospital, Créteil
  - Edouard Herriot Hospital, Lyon
  - Institut Paoli Calmette, Marseille
  - Nantes University Hospital, Nantes
  - Saint Louis Hospital, Paris
  - St Antoine, Paris
  - Haut-Leveque Hospital, Pessac
  - CHU de Poitiers, Poitiers
  - Purpan Hospital, Toulouse